CLINICAL TRIAL: NCT00407043
Title: A Prospective, Multicenter, Randomized Controlled Study of the Effect of Lotepredol Etabonate on The Initiation of Dry Eye Treatment With Topical Cyclosporine
Brief Title: Multicenter, Randomized, Controlled Study of the Effect of Lotemax on Initiation of Dry Eye Treatment With Restasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ophthalmic Consultants of Long Island (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Dr. Eric Donnenfeld, OCLI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Donnenfeld Review 1
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Dry Eye Disease; Keratoconjunctivitis Sicca
Keywords: Dry Eye Disease; Lotemax; Restasis; Loteprednol; Cyclosporine
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Loteprednol Etabonate; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lotemax
Drug: Restasis

SUMMARY:
To evaluate the impact of Lotemax on the initiation of Restasis therapy in patients with dry eye.

It is hypothesized that the anti-inflammatory activity of Lotemax may help mitigate the stinging with cyclosporine administration and the dry eye signs and symptoms experienced during the initiation of therapy.

DETAILED DESCRIPTION:
Dry eye is an ocular surface disease that produces discomfort and irritation. Estimated prevalence ranges from 20 million people in the US being affected with mild to moderate dry eye, to as many as one out of every five Americans.

A growing body of evidence has associated ocular inflammation with the signs and symptoms of dry eye.

Restasis is indicated to increase tear production in patients whose tear production is presumed to be suppressed due to ocular inflammation associated with a condition called keratoconjunctivitis sicca. The relief of dry eye signs and symptoms with Restasis therapy is often delayed by 1 to 6 months from the initiation of therapy. Stinging on installation, particularly when initiating therapy, has been reported.

Lotemax, an ophthalmic corticosteroid, targets inflammation with a unique, site-active mechanism of action.Structural modifications associated with an ester ophthalmic steroid make Lotemax highly lipid soluble, enhancing penetration into cells and enabling Lotemax to exert anti-inflammatory activity within the eye. Lotemax is indicated for the treatment of steroid responsive inflammatory conditions associated with the palpebral and bulbar conjunctiva, cornea, and anterior segment of the globe.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30 and 80 inclusive.
* Has not worn contact lenses for at least 1 month prior to the study and agrees to not wear contact lenses during study.
* Oral medications stable 1 month prior to study.
* Oral medications anticipated to be stable during 60 day study.
* Patient is in generally good & stable overall health.
* Patient likely to comply with eye drop regimen, study guidelines & study visits.
* Corneal stain > 1+ or Conjunctival stain > 1+ or OSDI equal or > 5 or using regular artificial tears at least on average twice daily.
* Informed consent signed.

Exclusion Criteria:

* History of Stevens-Johnson Syndrome or Ocular Pemphigoid.
* Punctal plugs inserted or punctal cautery in the past 3 months.
* Intra-ocular surgery within 6 months or ocular laser surgery within 3 months.
* History of liver disease.
* Pregnant or lactating women.
* Severe clinical vitamin deficiencies or history of vitamin overdose.
* Highly variable vitamin intake.
* Unstable use of systemic or topical medications known to create dry eye.
* Corneal pathology, which could, of itself, cause an ocular surface disorder.
* Use of glaucoma medications, topical or oral.
* Unstable diabetes mellitus.
* Allergy or sensitivity to Lotemax, Restasis or the OTC Tear Supplement.
* Use of topical steroids or Restasis within the past 1 month.
* Use of other topical ocular agents other than tear replacements within the past 1 week.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Questionnnaire Results
Lissamine green staining
Fluorescein Staining
Schirmer testing

CONTACTS AND LOCATIONS:
Overall Officials: Maria Howard, Study Director — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Lynbrook, New York, United States

REFERENCES:
- [Derived] Sheppard JD, Donnenfeld ED, Holland EJ, Slonim CB, Solomon R, Solomon KD, McDonald MB, Perry HD, Lane SS, Pflugfelder SC, Samudre SS. Effect of loteprednol etabonate 0.5% on initiation of dry eye treatment with topical cyclosporine 0.05%. Eye Contact Lens. 2014 Sep;40(5):289-96. doi: 10.1097/ICL.0000000000000049. PMID 25083776